CLINICAL TRIAL: NCT02746276
Title: Pharmacokinetics of Antimicrobials and Carriage of Antimicrobial Resistance Amongst Hospitalised Children With Severe Acute Malnutrition
Brief Title: Optimising Antibiotic Treatment for Sick Malnourished Children
Acronym: FLACSAM-PK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: KEMRI-Wellcome Trust Collaborative Research Program (Other); Centre for Research in Therapeutic Sciences, Strathmore University, Nairobi Kenya (Unknown); University College, London (Other); Centre for Microbiology Research, Kenya Medical Research Institute (Unknown); Centre for Clinical Research, Kenya Medical Research Institute (Unknown)
Responsible Party: Principal Investigator, James Berkley, Professor, University of Oxford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXTREC 47-15; KEMRI/SERU/CGMR-C/023/3161 (Other: KEMRI Scientific and Ethics Review Unit)
Record Dates: First submitted 2016-04-04; First posted 2016-04-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Malnutrition
Keywords: malnutrition; antibiotics; antimicrobial resistance; pharmacokinetics
MeSH Terms: conditions — Malnutrition | interventions — Ceftriaxone; Metronidazole

STUDY DESIGN:
Intervention Model Description: Sparse sample pharmacokinetics study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceftriaxone and metronidazole (Other): Pharmacokinetic study of ceftriaxone and metronidazole in malnourished children
  Interventions: Drug: Ceftriaxone; Drug: Metronidazole

INTERVENTIONS:
Drug: Ceftriaxone — Ceftriaxone is active against a broad spectrum of gram positive and gram negative bacteria, including intracellular bacteria (e.g. Salmonellae, Staphylococci). Its antibacterial effect is dependent on time above the minimum inhibitory concentration(MIC). Ceftriaxone is highly protein-bound and elimination depends on glomerular filtration rate. In severely ill adults, elimination is highly variable. Alteration in plasma proteins, volume of distribution and renal function in sick severely malnourished children could significantly alter pharmacokinetics (PK). Despite several published studies on the PK of ceftriaxone in children, none have included severe malnutrition.
  Other Names: Rocephin
Drug: Metronidazole — Metronidazole is effective against Giardia, which is common amongst children with SAM; and against other anaerobic infections, including small bowel bacterial overgrowth and Clostridium difficile colitis. Small cohort studies suggest there may be benefits for nutritional recovery. However, metronidazole can cause nausea and anorexia, potentially impairing recovery from malnutrition and may also cause liver and neurological toxicity. Changes in body composition as well as metabolic and drug elimination mechanisms may alter the potential toxicity or effective dose.
  Other Names: Flagyl

SUMMARY:
Children with severe malnutrition who are admitted sick to hospitals have a high mortality, usually because of infection. All children with severe malnutrition admitted to hospitals are treated with antibiotics. However, policymakers are not sure that the current antibiotics are the most effective. It is possible that the antibiotics that are currently used as second-line should be used first. Finding this out will need a large trial comparing different antibiotics. To prepare for such a trial the investigators first want to make sure that the doses given are correct for malnourished children. The investigators also want to check whether malnourished children more commonly carry resistant bacteria in their feces than well-nourished children. The study is important because the types of antibiotics and the doses needed to fight infection may be different in malnourished children because of the changes in their body due to malnutrition and the types of bacteria present.

DETAILED DESCRIPTION:
Children with complicated severe acute malnutrition (SAM) admitted to hospital in sub-Saharan Africa have an inpatient case fatality of 10 to 20%. Because children with SAM may not exhibit the usual signs of infection, World Health Organization (WHO) guidelines recommend routine antibiotics. However this is based on "low quality evidence". There is evidence from Centre for Geographic Medical Research - Coast (CGMR-C), Kilifi and from other centres in Africa that bacterial resistance to the currently recommended first-line antibiotics (gentamicin plus ampicillin or penicillin) may be a problem. It is possible that because of frequent illness and antibiotic exposure, malnourished children may be more likely to have resistant bacteria. Some hospitals in Africa are already increasing use of ceftriaxone as a first-line treatment. However, this is not based on any data that ceftriaxone actually improves outcomes. Of concern is that ceftriaxone use may also lead to further problems with antimicrobial resistance, including inducing extended spectrum beta-lactamase (ESBL) and other classes of resistance.

A further area where evidence for policy is lacking is on the use of metronidazole in severely malnourished children. The WHO guidelines recommend "Metronidazole 7.5 mg/kg every 8 h for 7 days may be given in addition to broad-spectrum antibiotics; however, the efficacy of this treatment has not been established in clinical trials." Metronidazole is effective against Giardia, which is common amongst children with SAM; and against other anaerobic infections, including small bowel bacterial overgrowth and Clostridium difficile colitis. Small cohort studies suggest there may be benefits for nutritional recovery. In Jamaica, half of the children admitted for nutritional rehabilitation had evidence of small bowel anaerobic bacterial overgrowth and this was improved by metronidazole. However, metronidazole can cause nausea and anorexia, potentially impairing recovery from malnutrition and may also cause liver and neurological toxicity. One small study of metronidazole in children with SAM conducted in in Mexico reported significantly prolonged clearance in SAM, without symptomatic toxicity, but suggesting a dosing frequency reduction. Overall, very few pharmacokinetic studies have been done in malnourished children. Changes in body composition as well as metabolic and drug elimination mechanisms may alter the potential toxicity or effective dose.

The investigators are planning a large clinical trial to assess the efficacy of ceftriaxone and metronidazole on mortality, nutritional recovery and antimicrobial resistance in sick, severely malnourished children. This preparatory work aims to determine the pharmacokinetics of ceftriaxone and metronidazole in 80 severely malnourished children who are admitted to three hospitals in Kenya in order to ensure dosing for the main trial is safe and in the therapeutic range. The study will also determine the frequency of faecal carriage of antimicrobial resistant enteric bacteria at presentation to hospital and at discharge following exposure to antibiotics and the hospital environment, comparing 360 children with, and 360 children without severe malnutrition at three different hospitals. Clear data on the benefits, risks and pharmacokinetics of these antimicrobials will influence policy on case management and antimicrobial stewardship in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Severe acute malnutrition(SAM) defined as:

  * Children aged 6 to 59 months with kwashiorkor; or Mid-Upper Arm Circumference (MUAC) <11.5cm; or weight-for height Z score <-3;
  * Children aged 2 to 5 months with kwashiorkor; or MUAC <11cm; or weight-for height Z score <-3; and weight >2.5 kilograms(kg);
* Eligible to receive intravenous antibiotics according to current national guidelines

For faecal carriage: children aged 2 to 59 months with and without SAM (as defined above) who are admitted to hospital with a syndrome requiring antimicrobial treatment under current national guidelines.

Exclusion Criteria:

* Admitted as a transfer from another hospital.
* Known ceftriaxone or metronidazole administration within the previous 7 days (pharmacokinetics(PK) study only).
* Known allergy or contraindication to ceftriaxone or metronidazole (including penicillin allergy) (PK study only).
* A specific clinical indication for another class of antibiotic (PK study only).
* Concurrent participation in a clinical trial (PK study only).
* Attending clinician's judgement that the child is so severely ill that adequate communication about the study with the parent or legal guardian is not possible.
* Refusal of consent

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of ceftriaxone | 24 hours
  To determine the pharmacokinetics of intravenous ceftriaxone given at currently recommended dose and frequency amongst severely malnourished, sick children.
Trough level of metronidazole | 8, 24, 48 and 72 hours
  To determine the pharmacokinetics of oral metronidazole given at currently recommended dose and frequency amongst severely malnourished, sick children.

SECONDARY OUTCOMES:
Prevalence of faecal carriage of extended spectrum beta-lactamase (ESBL) | Through study completion, an average of 5 days
  To determine the frequency of faecal carriage of ESBL at admission to hospital and at discharge amongst children admitted with and without severe malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: James A Berkley, Paediatrics, Principal Investigator — KEMRI Wellcome Trust Research Programme and University of Oxford
Locations (1):
- KEMRI WT Clinical Trials Facility, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Yes. Data sharing will be considered by the investigators, then by applying to the Data Governance Committee at CGMR,C who will ensure that appropriate ethical approval is in place for any new analysis.

REFERENCES:
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Bejon P, Mohammed S, Mwangi I, Atkinson SH, Osier F, Peshu N, Newton CR, Maitland K, Berkley JA. Fraction of all hospital admissions and deaths attributable to malnutrition among children in rural Kenya. Am J Clin Nutr. 2008 Dec;88(6):1626-31. doi: 10.3945/ajcn.2008.26510. PMID 19064524
- [Background] Talbert A, Thuo N, Karisa J, Chesaro C, Ohuma E, Ignas J, Berkley JA, Toromo C, Atkinson S, Maitland K. Diarrhoea complicating severe acute malnutrition in Kenyan children: a prospective descriptive study of risk factors and outcome. PLoS One. 2012;7(6):e38321. doi: 10.1371/journal.pone.0038321. Epub 2012 Jun 4. PMID 22675542
- [Background] Heikens GT, Bunn J, Amadi B, Manary M, Chhagan M, Berkley JA, Rollins N, Kelly P, Adamczick C, Maitland K, Tomkins A; Blantyre Working Group. Case management of HIV-infected severely malnourished children: challenges in the area of highest prevalence. Lancet. 2008 Apr 12;371(9620):1305-7. doi: 10.1016/S0140-6736(08)60565-6. No abstract available. PMID 18406865
- [Background] Chimhuya S, Kambarami RA, Mujuru H. The levels of malnutrition and risk factors for mortality at Harare Central Hospital-Zimbabwe: an observation study. Cent Afr J Med. 2007 May-Aug;53(5-8):30-4. doi: 10.4314/cajm.v53i5-8.62612. PMID 20355679
- [Background] Fergusson P, Tomkins A. HIV prevalence and mortality among children undergoing treatment for severe acute malnutrition in sub-Saharan Africa: a systematic review and meta-analysis. Trans R Soc Trop Med Hyg. 2009 Jun;103(6):541-8. doi: 10.1016/j.trstmh.2008.10.029. Epub 2008 Dec 5. PMID 19058824
- [Background] Trehan I, Goldbach HS, LaGrone LN, Meuli GJ, Wang RJ, Maleta KM, Manary MJ. Antibiotics as part of the management of severe acute malnutrition. N Engl J Med. 2013 Jan 31;368(5):425-35. doi: 10.1056/NEJMoa1202851. PMID 23363496
- [Background] Berkley JA, Lowe BS, Mwangi I, Williams T, Bauni E, Mwarumba S, Ngetsa C, Slack MP, Njenga S, Hart CA, Maitland K, English M, Marsh K, Scott JA. Bacteremia among children admitted to a rural hospital in Kenya. N Engl J Med. 2005 Jan 6;352(1):39-47. doi: 10.1056/NEJMoa040275. PMID 15635111
- [Background] Tansarli GS, Poulikakos P, Kapaskelis A, Falagas ME. Proportion of extended-spectrum beta-lactamase (ESBL)-producing isolates among Enterobacteriaceae in Africa: evaluation of the evidence--systematic review. J Antimicrob Chemother. 2014 May;69(5):1177-84. doi: 10.1093/jac/dkt500. Epub 2014 Jan 6. PMID 24398340
- [Background] Babirekere-Iriso E, Musoke P, Kekitiinwa A. Bacteraemia in severely malnourished children in an HIV-endemic setting. Ann Trop Paediatr. 2006 Dec;26(4):319-28. doi: 10.1179/146532806X152845. PMID 17132297
- [Background] Acquah SE, Quaye L, Sagoe K, Ziem JB, Bromberger PI, Amponsem AA. Susceptibility of bacterial etiological agents to commonly-used antimicrobial agents in children with sepsis at the Tamale Teaching Hospital. BMC Infect Dis. 2013 Feb 18;13:89. doi: 10.1186/1471-2334-13-89. PMID 23419199
- [Background] Blomberg B, Manji KP, Urassa WK, Tamim BS, Mwakagile DS, Jureen R, Msangi V, Tellevik MG, Holberg-Petersen M, Harthug S, Maselle SY, Langeland N. Antimicrobial resistance predicts death in Tanzanian children with bloodstream infections: a prospective cohort study. BMC Infect Dis. 2007 May 22;7:43. doi: 10.1186/1471-2334-7-43. PMID 17519011
- [Background] Aiken AM, Mturi N, Njuguna P, Mohammed S, Berkley JA, Mwangi I, Mwarumba S, Kitsao BS, Lowe BS, Morpeth SC, Hall AJ, Khandawalla I, Scott JAG; Kilifi Bacteraemia Surveillance Group. Risk and causes of paediatric hospital-acquired bacteraemia in Kilifi District Hospital, Kenya: a prospective cohort study. Lancet. 2011 Dec 10;378(9808):2021-2027. doi: 10.1016/S0140-6736(11)61622-X. Epub 2011 Nov 29. PMID 22133536
- [Background] Garot D, Respaud R, Lanotte P, Simon N, Mercier E, Ehrmann S, Perrotin D, Dequin PF, Le Guellec C. Population pharmacokinetics of ceftriaxone in critically ill septic patients: a reappraisal. Br J Clin Pharmacol. 2011 Nov;72(5):758-67. doi: 10.1111/j.1365-2125.2011.04005.x. PMID 21545483
- [Background] Lazzerini M, Tickell D. Antibiotics in severely malnourished children: systematic review of efficacy, safety and pharmacokinetics. Bull World Health Organ. 2011 Aug 1;89(8):594-607. doi: 10.2471/BLT.10.084715. Epub 2011 May 20. PMID 21836758
- [Background] Woerther PL, Angebault C, Jacquier H, Hugede HC, Janssens AC, Sayadi S, El Mniai A, Armand-Lefevre L, Ruppe E, Barbier F, Raskine L, Page AL, de Rekeneire N, Andremont A. Massive increase, spread, and exchange of extended spectrum beta-lactamase-encoding genes among intestinal Enterobacteriaceae in hospitalized children with severe acute malnutrition in Niger. Clin Infect Dis. 2011 Oct;53(7):677-85. doi: 10.1093/cid/cir522. PMID 21890771
- [Background] Paterson DL. "Collateral damage" from cephalosporin or quinolone antibiotic therapy. Clin Infect Dis. 2004 May 15;38 Suppl 4:S341-5. doi: 10.1086/382690. PMID 15127367
- [Background] Jones KD, Hunten-Kirsch B, Laving AM, Munyi CW, Ngari M, Mikusa J, Mulongo MM, Odera D, Nassir HS, Timbwa M, Owino M, Fegan G, Murch SH, Sullivan PB, Warner JO, Berkley JA. Mesalazine in the initial management of severely acutely malnourished children with environmental enteric dysfunction: a pilot randomized controlled trial. BMC Med. 2014 Aug 14;12:133. doi: 10.1186/s12916-014-0133-2. PMID 25189855
- [Background] Ignatius R, Gahutu JB, Klotz C, Steininger C, Shyirambere C, Lyng M, Musemakweri A, Aebischer T, Martus P, Harms G, Mockenhaupt FP. High prevalence of Giardia duodenalis Assemblage B infection and association with underweight in Rwandan children. PLoS Negl Trop Dis. 2012;6(6):e1677. doi: 10.1371/journal.pntd.0001677. Epub 2012 Jun 12. PMID 22720102
- [Background] Heikens GT, Schofield WN, Christie CD, Gernay J, Dawson S. The Kingston Project. III. The effects of high energy supplement and metronidazole on malnourished children rehabilitated in the community: morbidity and growth. Eur J Clin Nutr. 1993 Mar;47(3):174-91. PMID 8458315
- [Background] Lares-Asseff I, Cravioto J, Santiago P, Perez-Ortiz B. A new dosing regimen for metronidazole in malnourished children. Scand J Infect Dis. 1993;25(1):115-21. PMID 8460335
- [Background] Ribbing J, Jonsson EN. Power, selection bias and predictive performance of the Population Pharmacokinetic Covariate Model. J Pharmacokinet Pharmacodyn. 2004 Apr;31(2):109-34. doi: 10.1023/b:jopa.0000034404.86036.72. PMID 15379381
- See also: World Health Organization (2013) Pocket Book of Hospital Care for Children. Geneva. — http://apps.who.int/iris/bitstream/10665/81170/1/9789241548373_eng.pdf